CLINICAL TRIAL: NCT06333691
Title: Comparative Study Between Calcium Gluconate With Diosmin, Cabergoline and Cabergoline With Diosmin in Prevention of Ovarian Hyperstimulation Syndrome in High-risk Women Undergoing Intracytoplasmic Sperm Injection (ICSI) Procedures
Brief Title: Comparative Study Between Calcium Gluconate With Diosmin, Cabergoline and Cabergoline With Diosmin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Aya Mohammed Abdallah, Assistant lecturer in Clinical Pharmacy department, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Aya Mohammed
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: Calcium gluconate; Diosmin; Cabergoline; ICSI
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Calcium Gluconate; Cabergoline; Diosmin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): About 60 women patients,in which took IV infusion of calcium gluconate (Calcionate 10ml of 10% calcium gluconate, Memphis) in 200ml saline within 30 minutes of ovum pickup and contained for the next 3 days in addition to diosmin 2 tablets (500mg) t.d.s for 2 weeks.
  Interventions: Drug: Calcium Gluconate
- Group B (Active Comparator): About 60 women patients,in which took cabergoline (Dostinex 0.5 mg, Pfizer, Montreal, Canada) orally daily for 8 days after hCG triggering.
  Interventions: Drug: Calcium Gluconate
- Group C (Active Comparator): About 60 women patients,in which took diosmin , 2 tablets (500mg) t.d.s for 2 weeks in addition to cabergoline 1 tablet 0.5 mg/day orally for 8 days starting at the day of hCG injection.
  Interventions: Drug: Calcium Gluconate

INTERVENTIONS:
Drug: Calcium Gluconate — to compare the effectiveness of calcium gluconate, cabergoline and diosmin in preventing ovarian hyperstimulation syndrome in high-risk patient undergoing ICSI procedure.
  Other Names: Cabergoline; Diosmin

SUMMARY:
Ovarian hyperstimulation syndrome is a potentially fatal iatrogenic condition. This syndrome is characterized by a sudden increase of the vascular permeability which results in the development of a massive extravascular exudate in the peritoneal cavity, pleural, pericardium causing ascites, pleural and pericardial effusion.

Severe forms are also accompanied by electrolyte disturbances and cardiopulmonary, hepatic, renal, and hemoconcentration associated with increased thromboembolic risk.

This syndrome is avoidable by the judicious use of gonadotropins and careful monitoring of stimulation regimens.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome is a potentially fatal iatrogenic condition.

The major step to prevent hyperstimulation syndrome is to determine high risk patients as presence of polycystic ovarian syndrome, younger women with greater ovarian responsiveness, use of super active GnRH agonists, development of multiple immature and intermediate follicle during treatment, exposure to LH/hCG and previous history of hyperstimulation syndrome.

In addition, many different preventive modalities have been attempted such as decreasing the dose of FSH, using minimal or mild stimulating protocol as GnRH antagonists, use of insulin sensitizing agent as metformin, reduction the use of all follicles, decreasing the dose of hCG and administration of drugs which decrease capillary permeability as cabergoline, calcium gluconate, albumin, letrozole, hydroxyethyl starch and glucocorticoids.

Several different drugs have been used for prevention of hyperstimulation syndromes.

These include albumin, hydroxyethyl starch, aspirin, calcium, cabergoline, letrozole, and glucocorticoids. However, there is insufficient evidence about the benefits of these drugs in preventing hyperstimulation syndrome. Dopamine agonists (cabergoline) and calcium gluconate infusion are the most widely used preventive drugs.

Although these drugs have comparable effectiveness in preventing hyperstimulation syndrome with fewer maternal side effects, calcium maybe associated with arrhythmia

Recently attention has been focused on the use of Diosmin as a potent venotonic agent that decrease vascular permeability by reducing the release of inflammatory mediator such as prostaglandin E2 and thromboxane.

A study found that the combined use of diosmin and cabergoline in high-risk women undergoing ART was competent in avoiding hyperstimulation syndrome than using cabergoline alone. Moreover, this combination does not affect pregnancy rate, miscarriage nor multiple pregnancy

ELIGIBILITY:
Inclusion Criteria:

* High risk patient for OHSS is defined as previous history of OHSS or > 24 antral follicles of the ovaries on base line ultrasound (polycystic ovary)
* During ovarian stimulation-increased number of small follicles (8-12 mm)
* High AMH
* Rapidly rising serum E2
* High serum E2 at hCG trigger (>3000 pg/ ml) or presence of > 20 follicles on the day of retrieval, by ultrasound examination or >20 oocytes retrieved

Exclusion Criteria:

* patients with endocrine disorder e.g diabetes mellitus, Cushing's disease, and congenital adrenal hyperplasia,
* Patients with hypertension,
* Patients systemic disease e.g asthma, collagen vascular disease, hypercholesterolemia and sickle cell anemia.

Ages: 23 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
the incidence rate of moderate to severe OHSS. | 3 months
  OHSS is mainly characterized by abdominal distension, nausea, vomiting, diarrhea, hydrothorax, blood clotting disorders, and abnormal kidney function. Secondary outcomes included the clinical pregnancy rate, miscarriage rate, and live birth rate.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Sarhan, Professor, Study Chair — Professor of Pharmaceutics, Faculty of Pharmacy, Minia University.
Locations (1):
- Minia University, Faculty of Pharmacy, Minya, Egypt

REFERENCES:
- [Derived] Abdallah AM, Hussien AK, Alarfaj SJ, Elmasry TA, Kamal M, Sarhan H, Mosbeh MH, Sadek EM. Comparative study between calcium gluconate with diosmin, cabergoline, and cabergoline with diosmin in prevention of ovarian hyperstimulation syndrome in high-risk women undergoing intracytoplasmic sperm injection (ICSI) procedures. Front Pharmacol. 2025 Oct 27;16:1655866. doi: 10.3389/fphar.2025.1655866. eCollection 2025. PMID 41221041